CLINICAL TRIAL: NCT07318766
Title: Effect of Incentive Spirometer on Arterial Blood Gases in Liver Transplant Recipients
Brief Title: Incentive Spirometer in Liver Transplant Recipients
Acronym: LT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Collaborators: El-Sahel Teaching Hospital (Other Government); National Hepatology & Tropical Medicine Research Institute (Other Government)
Responsible Party: Principal Investigator, Aya Mohammed Abdel Magid Abdel Hamid, Lecturer of Clinical Pharmacy, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HS000132
Record Dates: First submitted 2025-12-07; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Liver Transplant Disorder
Keywords: Liver Transplant; Incentive Spirometer; Arterial Blood Gas

STUDY DESIGN:
Intervention Model Description: open label, parallel, prospective, randomized study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- mobilization and breathing exercises alone (No Intervention): Patients in the control group received standard post-transplant mobilization and breathing exercises as per institutional protocol. This included early mobilization, active limb exercises, and deep breathing exercises without the use of an intensive spirometry (IS) device. The exercise regimen was initiated on the first post-operative day and continued throughout the hospital stay.
- Incentive Spirometery plus standard exercises (Active Comparator): Patients in the intervention group received structured training on Incentive spirometry (IS) use commencing on the first post-operative day. A tri-flow volumetric IS device was utilized
  Interventions: Device: Incentive Spirometry

INTERVENTIONS:
Device: Incentive Spirometry — An intensive spirometry (IS) is a device that measures inhaled air volume and provides visual feedback as a piston rises during inspiration. It is widely used in respiratory and physical therapy to encourage slow, deep breathing, which helps expand the lungs, open airways, and mimic the natural deep breaths seen in yawning or sighing.
  Arms: Incentive Spirometery plus standard exercises

SUMMARY:
This study evaluated the effect of adjunctive incentive spirometer on arterial blood gases (ABGs) and early postoperative recovery in liver transplant recipients.

DETAILED DESCRIPTION:
In this prospective , randomized study, 40 adults undergoing living-donor liver transplantation (LT) were assigned to standard post-transplant mobilization and breathing exercises alone (n=20) or standard exercises plus structured IS training (n=20). Arterial blood gases ABG parameters (pH, PO₂, PCO₂, HCO₃-, SpO₂) were measured at baseline and on postoperative days 1-3. Linear mixed-effects models assessed group differences in ABG trajectories; slope analyses quantified decline and recovery phases. Secondary outcomes included intensive care unit (ICU) and hospital length of stay (LOS) and Post-operative pulmonary complications incidence.

ELIGIBILITY:
Inclusion Criteria:

1. age between 18 and 65 years,
2. scheduled to undergo Living Donor Liver Transplant (LDLT) as recipients
3. able to understand and follow instructions for incentive spirometry use

Exclusion Criteria:

1. multiorgan transplantation
2. moderate-to-severe pleural effusion at baseline
3. persistent elevation in renal function tests
4. history of bleeding esophageal varices within the preceding month
5. multicentric hepatocellular carcinoma (HCC)
6. active smoking
7. decompensated cardiac disease
8. alcoholic hepatitis as the primary etiology
9. cognitive impairment or blindness precluding participation in the rehabilitation protocol.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-11-01 (Actual); Study Completion 2025-11-01 (Actual)

PRIMARY OUTCOMES:
Arterial blood gas (ABG) parameters | 3 days (assessed at four time points: baseline (within 48 hours before surgery) and on post-operative days 1, 2, and 3)
  Arterial pH
Arterial Blood Gas (ABG) parameters | 3 days (assessed at four time points: baseline (within 48 hours before surgery) and at day 1,2, and 3 post-surgery)
  (2) partial pressure of carbon dioxide (PCO2, mmHg)
Arterial Blood Gas (ABG) parameters | 3 days (assessed at four time points: baseline (within 48 hours before surgery) and at day 1, 2, and 3 post-surgery)
  (3) Partial pressure of oxygen (PO2, mmHg)
Arterial Blood Gas (ABG) Parameters | 3 days (assessed at four time points: baseline (within 48 hours before surgery) and at day 1, 2, and 3 post-surgery)
  (4) bicarbonate concentration (HCO3-, mEq/L)
Arterial Blood Gas (ABG) Parameters | 3 days (assessed at four time points: baseline (within 48 hours before surgery) and at day 1, 2, and 3 post-surgery)
  (5) Oxygen saturation (SpO2, %).

SECONDARY OUTCOMES:
length of intensive care unit (ICU) stay | Perioperative period (Hospital stay duration)
  The length of intensive care unit (ICU) stay (days)
hospital stay | Perioperative period (Hospital Stay duration)
  total length of hospital stay (days)

CONTACTS AND LOCATIONS:
Overall Officials: Mona A. Abdulmohsen, MD, Principal Investigator — El-Sahel Teaching Hospital
Locations (1):
- El Sahel Teaching hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No